## Effectiveness of a Culturally Adapted Cognitive Behavioral Intervention to Reduce Psychological Distress and Improving Well-Being Among University Students During the COVID-19 Pandemic

[NCT ID not yet assigned] 21.03.2021

## **Informed Consent**

## Information about the project:

You are kindly invited to participate in our project, called "Effectiveness of a Culturally Adapted Cognitive Behavioral Intervention to Reducing Psychological Distress and Improving Well-Being Among University Students During the COVID-19 Pandemic" (2020.465.IRB3.184), led by Dr. Ceren Acartürk from the Department of Psychology at Koç University. Purpose of this project is to provide an online culturally adapted cognitive behavioral intervention (CA-CBI) to the university students who experience psychological distress during the COVID-19 pandemic. In scope of our project, the CA-CBI will be adapted to the university students and the problems they experience during the pandemic. After the adaptation process is completed, eligible participants will be randomly assigned to either intervention or control group. The participants in the intervention group will receive a 8-session CA-CBI in an online group format and the control group will be able to receive this intervention after the measurements are competed.

## Information about the questionnaire:

This part of the project aims to decide whether you are eligible to be invited to the intervention or not. Your participation in this study is entirely voluntary In case you accept to participate in the study, we will ask you to fill in an online survey, which will take approximately 10 minutes. After assessing your eligibility to receive the intervention, psychologists from our research team will contact you for the eight-week-intervention program.

Participation in this study is entirely upon your free will, without any coercion or obligation, your voluntary participation is essential. After deciding to participate, you may terminate the study without providing any specific reason at any time.

Under any circumstances expect one, the information you provide during the survey will not be matched with your credentials. The only exception is that you have an imminent suicide risk. In this case, a member of our team will reach you and make a referral after having an interview with you. Except this condition, all information you provide will only be used by the research team for academic purposes. The information you give will be kept in an encrypted database in which only the research team may have access. The information you provided will be recycled once the study is completed in an untraceable manner.

For your questions and comments, you may contact the responsible researchers: Assoc. Prof. Ceren Acartürk; cacarturk@ku.edu.tr

- I understood the information provided above and my questions are answered to my satisfaction. Without prejudice to my rights to terminate the study at any point, I agree to the conditions specified below and to participate in the study.
- I agree that the psychologists working with the research team will contact me in case of imminent suicide risk via my phone number.
- I know that my personal information will be recycled in an untraceable manner if my participation in the intervention program is not found eligible.
- I agree to participate in the study.
- I do not agree to participate in the study.